CLINICAL TRIAL: NCT06634849
Title: A Modular, Open Label, Dose Finding, Phase 1/2 Clinical Trial in Patients With Solid Tumours to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of PTT-4256.
Brief Title: An Open Label Dose Finding Study of PTT-4256 in Patients With Solid Tumours (RAISIC-1).
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pathios Therapeutics Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTT-4256-01
Record Dates: First submitted 2024-09-20; First posted 2024-10-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: PTT-4256, GPR65, oncology, cancer, RAISIC-1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTT-4256 (Experimental): Oral administration of PTT-4256 tablet with water
  Interventions: Drug: PTT-4256

INTERVENTIONS:
Drug: PTT-4256 — Single oral intake of PTT-4256 followed by treatment-free period of 3 days to assess safety, PK and PD. After 72-hr post dose PK sample, first 21day cycle of once daily PTT-4256 will begin to assess DLTs. Cohorts A1-A5 will receive 10mg, 20mg, 40mg, 80mg & 160mg. Following review by SRC, Cohort A6 participants will receive 300mg PTT-4256 daily.

SUMMARY:
This open label, dose escalation module will evaluate the safety, tolerability, PK, PD, and preliminary efficacy of PTT-4256 in participants with solid tumours using a combination of accelerated dose titration (ADT) and Bayesian Optimal Interval (BOIN) design.

DETAILED DESCRIPTION:
Module A - This module also aims to determine the MTD, if reached, and preliminary OBD (optimal biological dose) and RP2D (Recommended Phase 2 Dose). Eligible participants will be adults with cytologically or histologically confirmed solid malignancy and locally advanced or metastatic disease who require systemic treatment for their tumour and are either refractory to, have progressed on, are intolerant to, or are not otherwise a candidate, in the opinion of the Investigator, for any of the currently available standard treatments.

Module A will employ an ADT design for the first 2 cohorts (Cohorts A1 and A2) followed by a BOIN design for the subsequent cohorts (Cohorts A3 onwards). Participants will undergo a Screening period beginning up to 28 days prior to first dose and will be required to sign an informed consent form (ICF) before undertaking any study-specific procedures or assessments.

Participants who meet all of the inclusion and none of the exclusion criteria will be enrolled.

Safety oversight will be provided by a Safety Review Committee (SRC) comprising the Investigators, the Sponsor's Medical Monitor (MM)/representatives and other independent specialists (e.g. statistician).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of consent.
2. Participant has given written informed consent to participate in the study and is able and willing to adhere to the study protocol.
3. Participant has cytologically or histologically confirmed solid malignancy and has locally advanced or metastatic disease. Melanoma, non-small cell lung cancer, renal cell carcinoma, metastatic castrate-resistant prostate cancer, cervix cancer, triple negative breast cancer, colorectal cancer, gastric cancer are preferred solid tumours.
4. Participant must require systemic treatment for their tumour and either:

   1. be refractory to,
   2. have progressed on,
   3. be intolerant to, or
   4. be not otherwise a candidate - in the opinion of the Investigator - for any of the currently available standard treatments.
5. Participant has measurable disease per RECIST v1.1. Participants with non-measurable disease per RECIST v1.1 might be considered eligible upon discussion with the Sponsor.
6. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Participant has an estimated life expectancy of at least 3 months in the opinion of the Investigator.
8. Adequate haematological (blood or platelet transfusion not allowed within 7 days prior to Screening), liver, and renal function defined below (repeat measurement of borderline values permitted):

   * Haemoglobin ≥ 8.5 g/dL,
   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L,
   * Platelet count ≥ 90 x 109/L,
   * Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN), (or where ≤ 2 × ULN with known hepatobiliary metastases or Gilbert's syndrome),
   * Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 2.5 × ULN (or ≤ 5 ×ULN if liver metastases are present),
   * Estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m2 (calculated using Cockcroft-Gault).
9. Females:

   1. must not be pregnant or lactating, and must use acceptable, highly effective contraception from Screening until 90 days after last IMP administration. Effective forms of contraception are defined in Section 7.3.2,
   2. Females with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle,
   3. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study. WOCBP must not donate ova from signing informed consent until at least 90 days after the last IMP administration.
   4. Women of non-childbearing potential (WONCBP) must be postmenopausal for ≥12 months or ≥ 60 years of age at the time of consent (postmenopausal status is to be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L (except for participants on hormone replacement therapy) at Screening for amenorrhoeic female participants).
10. Males:

    1. must be surgically sterile (> 6 months since vasectomy with confirmation of no viable sperm),
    2. or if engaged in sexual relations (intercourse) with a WOCBP, either his partner must be surgically sterile (eg, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or an acceptable, highly effective contraceptive method must be used from Screening until 90 days after last IMP administration,
    3. Males with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle,
    4. Males must not donate sperm from the first dose of IMP until at least 90 days after the last dose of IMP

Exclusion Criteria:

1. Inability or unwillingness to adhere to the study protocol, including study procedures and oral intake of the IP.
2. Active primary central nervous system (CNS) malignancy, active CNS metastases or leptomeningeal disease. Participants with previously treated primary CNS malignancy or CNS metastases are eligible to participate if:

   1. they have stable and controlled neurological symptoms without deterioration;
   2. they have stable disease as assessed by imaging (preferably contrast-enhanced MRI) for at least 28 days prior to first IMP administration;
   3. they have no evidence of new or enlarging brain metastases; and
   4. they are not using corticosteroids for at least 7 days prior to first IMP administration.
3. Unresolved or unstable serious toxic side effects of prior chemotherapy or radiotherapy, ie, ≥ Grade 2 per CTCAE v5.0 except fatigue, alopecia, infertility, or those relating to palliative radiotherapy within 6 weeks prior to first IMP administration. Participants with residual AEs > Grade 1 considered not clinically significant may be considered eligible on a case-by-case basis, in discussion with the Sponsor.
4. Concurrent active or previous history of other malignancy within the past 2 years before first IMP administration except:

   1. Malignancy (other than in situ) treated with curative intent and with no known active disease present for ≥ 2 years before first IMP administration and felt to be at low risk of recurrence by the Investigator;
   2. Adequately treated non-melanoma skin cancer or lentigo malignant with no evidence of disease;
   3. Adequately treated in situ cancer without evidence of disease.
5. Received anti-cancer therapy (including chemotherapy, immunotherapy, radiation therapy, biologic therapy, or any investigational therapy) within 28 days or 5 half-lives of the therapeutic agent, whichever is shorter, prior to the first IMP administration. Palliative adiotherapy given within 28 days prior to the first IMP administration may be considered eligible on a case-by-case basis, in discussion with the Sponsor.
6. Uncontrolled symptomatic malignant effusion(s) or those requiring recurrent drainage in the opinion of the Investigator.
7. Participants with clinically significant active autoimmune or chronic inflammatory disease that is not well controlled with standard therapy in the opinion of the Investigator.
8. Grade 3 or higher immunotherapy-induced autoimmune hepatitis.
9. Participants with:

   1. symptomatic colitis of any CTCAE v5.0 Grade and aetiology within 4 weeks before first dosing,
   2. a history of autoimmune (including but not restricted to Crohn's disease, ulcerative colitis, and celiac's disease) or idiopathic (including but not restricted to pseudomembranous, ischaemic and microscopic) colitis, and/or,
   3. a history of drug-induced colitis of CTCAE v5.0 Grade 3 or higher.
10. History of primary immunodeficiency, bone marrow transplantation or solid organ transplantation.
11. Use of systemic immunosuppressive medication (including > 10 mg prednisolone per day or equivalent) within 14 days prior to the first IMP administration. Note that use of immunosuppressive medications as prophylaxis in participants with contrast allergies is acceptable. Adrenal replacement corticosteroid doses ≤10 mg daily prednisone equivalent are permitted, as are topical, inhaled, intra-articular or intra-nasal corticosteroids.
12. Participants with active Hepatitis B virus (HBV) hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at Screening) or Hepatitis C virus (HCV) hepatitis. Participants with resolved past HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
13. Participants with active HIV infection or known history of HIV infection.
14. Active infection requiring systemic antibacterial, antiviral or anti-fungal therapy for ≤ 7 days of first IMP administration. Note that participants on antibacterial, anti-fungal or antiviral prophylaxis are eligible.
15. Uncontrolled or recent history of clinically significant cardiovascular disease: Symptomatic heart failure (New York Heart Association classes II-IV), unstable angina, myocardial infarction, serious/uncontrolled/unstable cardiac arrhythmia, cerebral vascular accident, coronary/peripheral artery bypass graft surgery, transient ischaemic attack, or pulmonary embolism within 4 months prior to first IMP administration. Note that participants with small pulmonary emboli not thought to put them at higher risk may be considered eligible on a case-by-case basis, in discussion with the Sponsor.
16. Confirmed Baseline QTcF > 450 msec for males and > 470 msec for females (triplicate ECG) or history of torsades de pointes or history of congenital long QT syndrome. Note that participants with an apparent prolonged QT due to bundle branch block may be considered eligible on a case-by-case basis, in discussion with the MM.
17. History of clinically significant interstitial lung disease, or active non-infectious pneumonitis, or which may interfere with the detection or management of suspected drug related pulmonary toxicity.
18. Has had or is scheduled to have major surgery < 28 days prior to the first IMP administration. Elective surgical procedures not considered to put participants at higher risk of AEs may be allowed on a case-by-case basis, in discussion with the Sponsor.
19. Any other concurrent severe and/or uncontrolled medical, surgical or psychiatric and/or social condition which, in the view of the Investigator, could compromise the participant's safety or ability to participate in the study and make them unsuitable for participation.
20. Use of other investigational medicinal products within 2 weeks or at least 5 half-lives (whichever is longer) before IMP administration.
21. Must not have had a live vaccine administration ≤ 28 days prior to the first dose of the IMP.
22. Participants with known active or suspected alcohol or drug abuse that may interfere with the study in the opinion of the Investigator.
23. Gastrointestinal conditions that may affect oral absorption of drugs in the opinion of the Investigator, including but not restricted to gastroparesis and short bowel syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment emergent adverse events (TEAEs), Adverse events and Serious Adverse events as assessed by CTCAE V5.0 | First dose IMP to 21 to 28 days after last IMP dose.

SECONDARY OUTCOMES:
To determine the maximum tolerated dose (MTD) | Baseline to 21 to 28 days after last IMP dose.
  Determined by dose limiting toxicities (DLT) occurring in 21 days following initiation of once daily administration
To determine OBD | Baseline to 21 to 28 days after last IMP dose.
  Determined by dose limiting toxicities (DLT) occurring in 21 days following initiation of once daily administration and by SRC (safety review committee)
To determine R2PD | Baseline to 21 to 28 days after last IMP dose.
  Determined by dose limiting toxicities (DLT) occurring in 21 days following initiation of once daily administration and by SRC (safety review committee)
Plasma pharmacokinetics at single dose- Maximum observed concentration (Cmax) | Pre-dose, 2hours, 4hours, 8hours, and 12 hours Day 1, then at 24hours (Day2), 48 hours (Day 3) and 72 hours (Day4)
Plasma pharmacokinetics at single dose- Time to maximum concentration (Tmax) | Pre-dose, 2hours, 4hours, 8hours, and 12 hours Day 1, then at 24hours (Day2), 48 hours (Day 3) and 72 hours (Day4)
Plasma pharmacokinetics at single dose- Area under the drug concentration-time curve, from time zero extrapolated to infinity (AUC0-last) | Pre-dose, 2hours, 4hours, 8hours, and 12 hours Day 1, then at 24hours (Day2), 48 hours (Day 3) and 72 hours (Day4)
Plasma pharmacokinetics at single dose- Area under curve from zero to 24hrs (AUC0-24) | Pre-dose, 2hours, 4hours, 8hours, and 12 hours Day 1, then at 24hours (Day2), 48 hours (Day 3) and 72 hours (Day4)
Plasma pharmacokinetics at single dose- Apparent terminal half-life (t1/2) | Pre-dose, 2hours, 4hours, 8hours, and 12 hours Day 1, then at 24hours (Day2), 48 hours (Day 3) and 72 hours (Day4)
Plasma PK at steady state- Maximum observed concentration in the dosing interval at steady state (Cmax,ss) | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- Minimum observed concentration in the dosing interval at steady state (Cmin,ss) | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- Average steady state concentration (Cavg,ss) | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- e to maximum observed plasma analyte concentration at steady state (Tmax,ss) | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- Time to minimum concentration at steady state (Tmin,ss) | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- Areas under the drug concentration-time curve over a dosing interval using the 'the linear up and log down' method (AUC0-tau) | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- Swing | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- Fluctuation | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- Trough concentration (Ctrough) | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- accumulation ratios (RA) of Cmax | Baseline to Cycle 2 Day 2 - 22 days
Plasma PK at steady state- accumulation ratios (RA) of Area under curve (AUC) | Baseline to Cycle 2 Day 2 - 22 days

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Blacktown Hospital, Blacktown, New South Wales
  - Scientia Clinical Research, Randwick, New South Wales
  - Southern Oncology Clinical Research Unit (SOCRU), Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No